CLINICAL TRIAL: NCT02967120
Title: A Multicentral Prospective Study on Prediction of Malignant Progression of Oral Epithelial Dysplasia With p16 Hydroxymethylation
Brief Title: Early Diagnosis of Oral Cancer by Detecting p16 Hydroxymethylation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Municipal Administration of Hospitals (Other Government)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Zhaojun Liu, PhD, Beijing Municipal Administration of Hospitals
Other Study IDs: XM201303
Record Dates: First submitted 2016-11-16; First posted 2016-11-17 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Oral Epithelial Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral mucosal biopsy tissues were formalin fixed , paraffin embedded , sliced；or frozen tissues;
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- p16 hydroxymethylation status: patients with p16 hydroxymethylation
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The purpose of this study is to verify the function of p16 hydroxymethylation diagnostic reagents in early diagnosis of oral cancer.

DETAILED DESCRIPTION:
Background:Oral epithelial dysplasia (OED) is one of the common precancerous lesions among Chinese adults. To investigate the clinical predictive value of p16 hydroxymethylation diagnostic reagents in the early diagnosis of oral cancer, the investigators carried out the prospective multi-center double-blind cohort study.

Methods:265 patients with histologically confirmed mild or moderate OED were included in the present study. After the bisulfite modification and tet assistant bisulfite modification, MethyLight and Methylation-specific PCR (MSP) assays were used to analyze p16 methylation and status in these patients. Building three follow-up queue by p16-methylated, p16-hydroxymethylation and p16-unmethylated. The Statistical analysis used SPSS16.0. All P-values were two-sided. P<0.05 was considered to test for statistical significance difference.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of oral lesions meet the epithelial diagnostic criteria for mild to moderate grade OED;
* No local area stimulate by residual root and crown, sharp cusp, poor restoration and biting cheek or lips;
* Without the treatment history by laser , radiation or chemical;
* Be able to Sign the informed consent;

Exclusion Criteria:

* Histopathological diagnosis of oral lesions do not meet the epithelium of mild to moderate dysplasia diagnostic criteria; histological diagnosis of severe grade OED or malignant disease;
* Pregnancy or breast-feeding women;
* Serious heart, lung, liver , kidney and other systemic diseases local area stimulate by residual root and crown, sharp cusp, poor restoration and biting cheek or lips;
* OED treatment history by LASER, radiotherapy, or chemotherapy;
* Tumor and psychiatric patients;
* Patients are unable to cooperate;

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 336 patients with mild or moderate oral epithelial dysplasia were selected. 145 of them are collected from Peking University of Stomatology and 165 were from Capital Medical University School of Stomatology and other 26 were from Fourth Military Medical University School of Stomatology.All of the patients with OED had been diagnosed pathologically by at least two senior pathologists using the criteria from '2005 WHO Classification System' and The oral tissue pathology diagnostic criteria (oral histopathology Edition Sixth).All cases involved primary lesions without any LASER, radiation therapy or chemotherapy.
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Cancer rate in patients with oral epithelial dysplasia containing or NOT containing p16 hydroxymethylation | from 3 months to 60 months
  Among these cases, oral specimens from 24 patients were p16-hydroxymethylation, 54 patients were p16-methylation and 187 patients were p16-unmethylation. The cancer rate in the p16-hydroxymethylation patients during the followup period will be compared with that in the other two groups.

SECONDARY OUTCOMES:
Disease free survival of patients with oral epithelial dysplasia containing or Not containing p16 hydroxymethylation | from 3 months and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Dajun Deng, MD, Study Director — Peking University Cancer Hosptial and Institute
Locations (1):
- Peking University Cancer Hosptial and Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The number of the participants of different groups and the followup information will be shared with other researchers after the end of the study.

REFERENCES:
- [Background] Liu H, Liu XW, Dong G, Zhou J, Liu Y, Gao Y, Liu XY, Gu L, Sun Z, Deng D. P16 Methylation as an Early Predictor for Cancer Development From Oral Epithelial Dysplasia: A Double-blind Multicentre Prospective Study. EBioMedicine. 2015 Mar 23;2(5):432-7. doi: 10.1016/j.ebiom.2015.03.015. eCollection 2015 May. PMID 26137587
- [Background] Cao J, Zhou J, Gao Y, Gu L, Meng H, Liu H, Deng D. Methylation of p16 CpG island associated with malignant progression of oral epithelial dysplasia: a prospective cohort study. Clin Cancer Res. 2009 Aug 15;15(16):5178-83. doi: 10.1158/1078-0432.CCR-09-0580. Epub 2009 Aug 11. PMID 19671846
- [Derived] Liu H, Liu Z, Liu XW, Xu S, Wang L, Liu Y, Zhou J, Gu L, Gao Y, Liu XY, Shi H, Sun Z, Deng D. A similar effect of P16 hydroxymethylation and true-methylation on the prediction of malignant transformation of oral epithelial dysplasia: observation from a prospective study. BMC Cancer. 2018 Sep 24;18(1):918. doi: 10.1186/s12885-018-4787-6. PMID 30249192